CLINICAL TRIAL: NCT06345950
Title: Pharmacokinetics and Safety of a New Micellar Glutathione Formulation in Human Participants
Brief Title: Pharmacokinetics and Safety of a New Micellar Glutathione Formulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Factors Group of Nutritional Companies Inc. (Industry)
Collaborators: Isura (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-04-003
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Bioavailability; Safety
Keywords: pharmacokinetics; glutathione; bioavailability; safety; micellar delivery system
MeSH Terms: interventions — glutathione pegylated liposomal doxorubicin

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to interventions in a crossover design to assess the pharmacokinetics over 24 hours; subsequently, the safety of one intervention with higher bioavailability is evaluated in an additional single-arm, 30-day trial.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Liposomal Glutathione (Experimental): Each participant receives their treatment i.e., Liposomal Glutathione hard gel capsules at a total dose of 500 mg glutathione. Treatments are consumed with a glass of water (approx. 125mL), followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at different time points up to 24 hours post-dose.
  A washout period of at least 14 days between each treatment is used.
  Interventions: Dietary Supplement: Liposomal Glutathione
- Standard Glutathione (Experimental): Each participant receives their treatment i.e., Standard Glutathione hard gel capsules at a total dose of 500 mg glutathione. Treatments are consumed with a glass of water (approx. 125mL), followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at different time points up to 24 hours post-dose.
  A washout period of at least 14 days between each treatment is used.
  Interventions: Dietary Supplement: Standard Glutathione
- New Micellar Glutathione (Lipomicel) (Experimental): Each participant receives their treatment i.e., LipoMicel Glutathione soft gel capsules at a total dose of 600 mg glutathione. Treatments are consumed with a glass of water (approx. 125mL), followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at different time points up to 24 hours post-dose.
  A washout period of at least 14 days between each treatment is used.
  Interventions: Dietary Supplement: New Micellar Glutathione (Lipomicel)

INTERVENTIONS:
Dietary Supplement: Liposomal Glutathione — A maximum single dose of 500 mg glutathione (hard gel capsules)
  Arms: Liposomal Glutathione
Dietary Supplement: Standard Glutathione — A maximum single dose of 500 mg glutathione (hard gel capsules)
  Arms: Standard Glutathione
Dietary Supplement: New Micellar Glutathione (Lipomicel) — A maximum single dose of 600 mg glutathione (soft gel capsules)
  Arms: New Micellar Glutathione (Lipomicel)

SUMMARY:
This study seeks to determine the short-term effects of daily oral supplementation with a new micellar Glutathione formulation (LipoMicel) on the oral absorption and safety of glutathione in healthy volunteers.

The primary objective of this study is to evaluate and compare the pharmacokinetics of a novel micellar Glutathione (GSH) formulation with that of a standard formulation as well as a liposomal GSH formulation. The secondary objective is to evaluate the safety of a new micellar GSH formulation with higher bioavailability in human participants over a 30-day study period.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 21-65 years
* healthy, good physical condition
* voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* use of anti-inflammatory or non-steroidal anti-inflammatory drugs
* previous history of cardiovascular disease or acute or chronic inflammatory disease
* use of antioxidant supplements or cholesterol-lowering agents
* change of diet habits or lifestyle (diet, physical activity, etc.)
* alcohol or substance abuse history
* use of nicotine or tobacco
* participation in another investigational study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
AUC: the area under the concentration-time curve | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested glutathione in healthy adult volunteers and compare the Area under the plasma concentration versus time curve (AUC) with that of other capsules containing glutathione.
Cmax: maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested glutathione in healthy adult volunteers and compare the peak plasma concentration (Cmax) with that of other capsules containing glutathione.
Tmax: the time point of maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested glutathione in healthy adult volunteers and compare the time point of maximum plasma concentration (Tmax) with that of other capsules containing glutathione.

SECONDARY OUTCOMES:
Alanine aminotransferase (ALT) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in liver function based on ALT.
Aspartate aminotransferase (AST) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in liver function based on AST.
Alkaline phosphatase (ALP) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in liver function based on ALP.
Bilirubin | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in liver function based on Bilirubin.
Serum creatinine | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in kidney function based on Serum creatinine.
Blood urea nitrogen (BUN) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in kidney function based on BUN.
Glomerular filtration rate (GFR) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in kidney function based on GFR.
C-reactive protein (CRP) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in inflammatory response based on CRP.
White blood cell count (WBC) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in complete blood count based on WBC.
Hemoglobin (Hb) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in complete blood count based on Hb.
Hematocrit (Hct) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in complete blood count based on Hct.
Platelet count | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in complete blood count based on Platelet count.
  .
Fasting blood glucose | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in blood glucose levels based on fasting blood glucose.
Total cholesterol | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in lipid profile based on total cholesterol.
Low-density lipoprotein (LDL) cholesterol | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in lipid profile based on LDL.
High-density lipoprotein (HDL) cholesterol | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in lipid profile based on HDL.
Triglycerides | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in lipid profile based on triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Solnier, PhD, Principal Investigator — Isura
Locations (1):
- ISURA, Burnaby, British Columbia, Canada